CLINICAL TRIAL: NCT06138041
Title: Effect of Intravenous Lidocaine Infusion on Postoperative Pulmonary Complications in Patients Undergoing Minimally Invasive Esophagectomy: a Double-center, Double-blind, Randomized Controlled Trial
Brief Title: Intravenous Lidocaine Infusion Reduce Postoperative Pulmonary Complications in Patients Undergoing Minimally Invasive Esophagectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yihao Zhu, Dr., Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: scchec-20231113
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pneumonia; Postoperative Pulmonary Atelectasis; Postoperative Pulmonary Edema
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Experimental): At the same time of induction of general anesthesia, an intravenous lidocaine bolus of 2mg/kg will be administered, followed by a continuous infusion of intravenous lidocaine at 2 mg/kg/h until the participate transfer out of postoperative anesthesia care unit.
  Interventions: Drug: intravenous lidocaine infusion
- control group (Placebo Comparator): The control group will receive the same volume of normal saline in bolus and continuous infusion.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: intravenous lidocaine infusion — Lidocaine bolus of 2mg/kg after induction , and then continuous infusion with 2 mg/kg/h until the participate transfer out of postoperative anesthesia care unit.
  Arms: lidocaine group
Drug: Saline — Same volume of normal saline in bolus and continuous infusion as lidocaine group.
  Arms: control group

SUMMARY:
The goal of this double-center, double-blind, randomized controlled clinical trial is to compare the effect of intravenous lidocaine infusion on postoperative pulmonary complications in patients undergoing minimally invasive esophagectomy. The main question it aims to answer are whether intravenous lidocaine reduce postoperative pulmonary complications in patients undergoing minimally invasive esophagectomy. Participants will be given intravenous lidocaine infusion in lidocaine group or placebo in control group.

ELIGIBILITY:
Inclusion Criteria:

Patients between 18 and 85 years of age with a recent schedule for MIE are screened for this study. Patients who show clear consciousness and ASA status I - III will be included as eligible participants.

Exclusion Criteria:

The exclusion criteria are as follows: patients with severe psychiatric disorders, such as schizophrenia, depression, dementia, etc.; severe hepatic insufficiency (concentration of glutamic oxaloacetic transaminase, glutamic pyruvic transaminase or bilirubin ≥2.5 times the upper limit of normal); renal impairment (creatinine clearance <60 mL/min); allergy to amide local anesthetics; history of seizures; presence of II/III atrioventricular block; patients with severe sinus bradycardia or sick sinus syndrome; patients with Adams-Stokes syndrome or pre-excitation syndrome; intracardiac block (e.g. complete bundle branch block, atrioventricular block); serum potassium ion concentration below 2.5 or above 5.0 mmol/L; PH>7.55 or PH<7.2. Patients will be discontinued if any of the following situations occur: the patient has an allergic reaction, severe cardiovascular events that cannot be managed with symptomatic treatment, and the patient is unwilling to continue the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of PPCs | 1, 2, 3, 4, 5, 6, 7 days after surgery
  Pulmonary complications is defined as one or more of the following complications: respiratory infection; respiratory failure; pneumothorax;atelectasis; pleural effusion; bronchospasm; aspiration pneumonitis; anastomotic fistula

SECONDARY OUTCOMES:
respiratory infection | 1, 2, 3, 4, 5, 6, 7 days after surgery
respiratory failure | 1, 2, 3, 4, 5, 6, 7 days after surgery
pneumothorax;atelectasis | 1, 2, 3, 4, 5, 6, 7 days after surgery
pleural effusion | 1, 2, 3, 4, 5, 6, 7 days after surgery
bronchospasm | 1, 2, 3, 4, 5, 6, 7 days after surgery
aspiration pneumonitis | 1, 2, 3, 4, 5, 6, 7 days after surgery
anastomotic fistula | 1, 2, 3, 4, 5, 6, 7 days after surgery
moderate to severe pain within 24 and 48 hours at rest and when coughing | 24 and 48 hours after surgery
moderate to severe pain within 24 and 48 hours at coughing | 24 and 48 hours after surgery
additional rescue analgesics use | 24 and 48 hours after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang F, Zhang H, Peng X, Liu M, Wang H, Song Y, Jia X, Zhu T, Zhu Y. Effect of intravenous lidocaine infusion on postoperative pulmonary complications in patients undergoing minimally invasive esophagectomy: a study protocol of double-center, double-blind, randomized controlled trial. Trials. 2025 Nov 11;26(1):490. doi: 10.1186/s13063-025-09213-x. PMID 41219803